CLINICAL TRIAL: NCT00882609
Title: 18F-Fluoride PET/CT Versus 99mTc-MDP Scanning for Detecting Bone Metastases: A Randomized, Multi-Center Trial to Compare Two Bone Imaging Techniques
Brief Title: F18PET/CT Versus TC-MDP Scanning to Detect Bone Mets
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: American College of Radiology - Image Metrix (Industry)
Collaborators: World Molecular Imaging Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: AMI-2008-01
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Bone Metastases
Keywords: bone metastasis; bone metastases; Sodium Fluoride; F18 Fluoride; bone scan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TC-MDP Bone Scan (Active Comparator): Patients without known bone metastases who are newly diagnosed with ≥ stage 3 breast cancer, ≥ stage 3 lung cancer, or ≥ stage 2 prostate cancer (and/or PSA >10 micrograms/L), including patient with recurrent breast, lung or prostate cancer; Patient is scheduled to undergo a conventional bone scan
  Interventions: Device: Bone Scan: F18-Fluoride PET/CT or TC-MDP
- F18-Fluoride PET/CT (Experimental): Patients without known bone metastases who are newly diagnosed with ≥ stage 3 breast cancer, ≥ stage 3 lung cancer, or ≥ stage 2 prostate cancer (and/or PSA >10 micrograms/L), including patient with recurrent breast, lung or prostate cancer; Patient is scheduled to undergo a conventional bone scan
  Interventions: Device: Bone Scan: F18-Fluoride PET/CT or TC-MDP

INTERVENTIONS:
Device: Bone Scan: F18-Fluoride PET/CT or TC-MDP — Each patient will be randomized into one of two groups with one group receiving Sodium Fluoride F18 Injection and the other receiving the control agent, 99mTc-MDPSodium Fluoride F18 Injection Dosing and Administration. The dose will be tailored for the specific patient for whom the dose was ordered. The dose of Sodium Fluoride F18 Injection administered will range from 5-10 mCi/patient.Each patient randomized to the control group will be administered 99mTc-MDP as a single intravenous bolus dose. The administered radioactivity will be determined based on the sites routine clinical practice for conventional bone imaging.

SUMMARY:
The primary objective is to compare the diagnostic performance of 18F- Fluoride PET/CT scanning to that of conventional bone scanning for detecting cancer that has spread to the bone (bone metastasis). The intent of the study is to determine whether 18F-Fluoride PET/CT will lead to improved treatment and patient outcomes.

DETAILED DESCRIPTION:
The trial will accrue four hundred-eighty eight (488) evaluable patients with breast cancer, prostate cancer or lung cancer (approximately 163 of each cancer type) referred for routine bone scanning by their respective physicians. The specific stages of cancer required for eligibility are described in the eligibility criteria.

Approximately eleven to fifteen qualified clinical centers will participate in the trial, with target enrollment for each site set at roughly 40-50 patients per site.

The images of the patients will be transmitted to ACR Image Metrix, an imaging contract research organization (iCRO), for quality assurance and archival. iCRO will conduct blinded core lab interpretations by 3 radiologists who have not been involved in the design of the trial nor the clinical image interpretation. The data from the core lab readings will be compared with the deliberations of a multidisciplinary panel of oncology experts who will be blinded to the initial scan results and will determine the standard of evidence (truth) for each patient. The analysis will be based on this comparison.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years old at the time of the drug administration (Patient may be male or female of any race / ethnicity.)
* Patient or patient's legally acceptable representative cognitively provides written informed consent
* Patients without known bone metastases who are newly diagnosed with ≥ stage 3 breast cancer, ≥ stage 3 lung cancer, or ≥ stage 2 prostate cancer (and/or PSA >10 micrograms/L), including patient with recurrent breast, lung or prostate cancer
* Patient is scheduled to undergo a conventional bone scan
* Patient is capable of complying with study procedures
* Patient is able to remain still for duration of imaging procedure (about one hour)
* Patient may have had a prior PET or PET/CT scan for staging/restaging.

Exclusion Criteria:

* Patient is < 18 years old at the time of the drug administration
* Patient is pregnant or nursing;

  * testing on site at the institution (urine or serum ßHCG) within 24 hours prior to the start of investigational product administration
  * obtaining surgical history (e.g., tubal ligation or hysterectomy)
  * confirming the subject is post menopausal, with a minimum 1 year without menses
* Patient has any other condition or personal circumstance that, in the judgment of the investigator, might interfere with the collection of complete good quality data
* Patient has known bone metastases
* Patient has previously received [18F]NaF in the last thirty days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Analysis of the diagnostic performance of [18F]NaF fluoride PET/CT scanning | 6 Months
  The primary endpoint will be an analysis of the diagnostic performance of [18F]NaF fluoride PET/CT scanning to that of conventional bone scanning for detecting cancer that has spread to the bone (bone metastasis). The hypothesis is that PET/CT is superior to conventional bone scanning for detecting bone metastases. The primary metrics used for comparison will be the relative areas under the ROC curves generated by blinded core lab interpretations of the scans.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Czernin, MD, Principal Investigator — World Molecular Imaging Society
Locations (19):
- United States (15):
  - Scottsdale Medical Imaging, Scottsdale, Arizona
  - Silicon Valley Imaging, Freemont, California
  - Cedar-Sinai Medical Center, Los Angeles, California
  - VA West Los Angles Medical Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - SouthCoast Imaging Center, Savannah, Georgia
  - University of Michigan Health System, Ann Arbor, Michigan
  - Saint Luke's Hospital, Kansas City, Missouri
  - John Cochran Veterans Administration, St Louis, Missouri
  - Saint Louis University, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - New York Presbyterian Weill Cornell, New York, New York
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
- Peter MacCallum, Melbourne, Victoria, Australia
- PET-CT Linz - St. Vicent's Hospital, Linz, Linz, Austria
- Hospitais da Universidade de Coimbra, Coimbra, Portugal, Portugal
- University Hospital Zurich, Zurich, Switzerland, Switzerland